CLINICAL TRIAL: NCT00974792
Title: A Phase II Single Arm Study of the Use of CODOX-M/IVAC With Rituximab (R-CODOX-M/IVAC) in the Treatment of Patients With Diffuse Large B-Cell Lymphoma (International Prognostic Index High or High-Intermediate Risk)
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With Diffuse Large B-Cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000644893; CRUK-UCL-R-CODOX-M/IVAC; EUDRACT-2005-003479-19; EU-20956
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-09

CONDITIONS: Lymphoma
Keywords: stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — pegfilgrastim; Rituximab; Cyclophosphamide; Cytarabine; Doxorubicin; etoposide phosphate; Ifosfamide; Leucovorin; Methotrexate; Vincristine

INTERVENTIONS:
Biological: pegfilgrastim
Biological: rituximab
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: etoposide phosphate
Drug: ifosfamide
Drug: leucovorin calcium
Drug: methotrexate
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cell-killing substances to them. Giving more than one drug (combination chemotherapy) together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with rituximab works in treating patients with diffuse large B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate in patients with high- or high/intermediate-risk diffuse large B-cell lymphoma treated with CODOX-M/IVAC comprising cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, methotrexate, ifosfamide, etoposide phosphate, and cytarabine with rituximab.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the progression-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV on days 1 and 11 and CODOX-M comprising doxorubicin hydrochloride IV on day 1, cyclophosphamide IV on days 1-5, vincristine sulfate IV on days 1 and 8, methotrexate IV over 12 hours on day 10, and leucovorin calcium IV or orally every 3-6 hours beginning 24-36 hours after methotrexate. Patients also receive CNS prophylaxis comprising cytarabine intrathecally (IT) on days 1 and 3 and methotrexate IT on day 15. Patients with high-risk disease receive an additional dose of cytarabine IT on day 5 and methotrexate IT on day 17. Patients also receive pegfilgrastim subcutaneously (SC) on day 11. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of CODOX-M course 1, patients receive rituximab IV on day 1** and IVAC comprising etoposide phosphate IV over 1 hour and ifosfamide IV over 1 hour on days 1-5, cytarabine IV over 3 hours (every 12 hours) on days 1 and 2, and methotrexate IT on day 5. Patients with high-risk disease receive cytarabine IT on days 7 and 9. Patients also receive pegfilgrastim SC on day 7. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

NOTE: **Patients with high-risk disease also receive rituximab IV on days 21 and 42 after day 1 of course 4 (IVAC).

Treatment with R-CODOX-M and R-IVAC repeats every 28 days alternatively for 2 courses each in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell non-Hodgkin lymphoma

  * International Prognostic Index (IPI) score high-intermediate (score = 3) OR high (score = 4 or 5), defined as:

    * Stage III or IV disease
    * Raised lactic dehydrogenase and poor performance status (WHO performance status 2-4)
  * All morphological variants included
  * B-cell nature of the proliferation must be verified by a positive anti-CD20 antibody (i.e., CD20-positive disease)
* No T-cell lymphoma
* No history of treated or non-treated indolent lymphoma

  * Patients newly diagnosed who have large B-cell lymphoma with some small cell infiltration in the bone marrow or lymph node may be allowed

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Life expectancy > 3 months
* ANC > 1,500/mm^3*
* Platelet count > 100,000/mm^3*
* Serum creatinine < 150 μmol/L*
* Serum bilirubin < 35 μmol/L*
* AST and/or ALT < 2.5 times upper limit of normal* NOTE: *Unless attributed to bone marrow infiltration by lymphoma.
* Fertile patients must use effective contraception
* Normal MUGA or echocardiogram without areas of abnormal contractility
* LVEF ≥ 50% and only tested if patient meets 1 of the following criteria:

  * History of diabetes
  * Prior cardiac disease, hypertension, or abnormal resting ECG
* No history of heart failure or uncontrolled angina pectoris
* No cardiac contraindication to doxorubicin hydrochloride (e.g., abnormal contractility on echocardiography or MUGA)
* No neurological contraindication to vincristine sulfate (e.g., pre-existing diabetic neuropathy)
* No concurrent uncontrolled medical condition
* No other serious active disease
* No general status that, according to the investigator, does not allow the administration of 2 courses of CODOX-M/IVAC
* No active malignant disease within the past 10 years except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix
* No positive serology for HIV or hepatitis B or C
* No medical or psychiatric conditions that compromise the patient's ability to give informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, radiotherapy, or other investigational drug for diffuse large B-cell non-Hodgkin lymphoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Complete response rate

SECONDARY OUTCOMES:
Toxicity
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: A. McMillan, Principal Investigator — Nottingham City Hospital
Locations (1):
- Nottingham City Hospital, Nottingham, England, United Kingdom

REFERENCES:
- [Derived] McMillan AK, Phillips EH, Kirkwood AA, Barrans S, Burton C, Rule S, Patmore R, Pettengell R, Ardeshna KM, Lawrie A, Montoto S, Paneesha S, Clifton-Hadley L, Linch DC. Favourable outcomes for high-risk diffuse large B-cell lymphoma (IPI 3-5) treated with front-line R-CODOX-M/R-IVAC chemotherapy: results of a phase 2 UK NCRI trial. Ann Oncol. 2020 Sep;31(9):1251-1259. doi: 10.1016/j.annonc.2020.05.016. Epub 2020 May 26. PMID 32464282